CLINICAL TRIAL: NCT05718258
Title: A Phase 1, Multi-center, Parallel, Open-label, Pharmacokinetic, Safety, and Tolerability Study of Venglustat Given as a Single Dose in Adult Participants With Mild, Moderate, and Severe Hepatic Impairment and in Matched Participants With Normal Hepatic Function
Brief Title: A Study in Adults to Investigate the Impact of Mild, Moderate, and Severe Hepatic Impairment on Pharmacokinetics of Venglustat Compared to Participants With Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: POP16551; U1111-1261-7500 (Registry Identifier: ICTRP); 2022-000945-34 (EudraCT Number)
Record Dates: First submitted 2023-01-30; First posted 2023-02-08 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Hepatic Function Abnormal
MeSH Terms: conditions — Liver Diseases | interventions — venglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Participants with mild hepatic impairment (Experimental): Venglustat single dose on Day 1
  Interventions: Drug: Venglustat (GZ402671)
- Participants with normal hepatic function (Experimental): Venglustat single dose on Day 1
  Interventions: Drug: Venglustat (GZ402671)
- Participants with moderate hepatic impairment (Experimental): Venglustat single dose on Day 1
  Interventions: Drug: Venglustat (GZ402671)
- Participants with severe hepatic impairment (Experimental): Venglustat single dose on Day 1
  Interventions: Drug: Venglustat (GZ402671)

INTERVENTIONS:
Drug: Venglustat (GZ402671) — Pharmaceutical form: tablet
  Route of administration: oral

SUMMARY:
This is a parallel, Phase 1, four arm, open-label, single dose, multicenter study to evaluate the impact of hepatic impairment on venglustat exposure following treatment with venglustat.

The purpose of this study is to assess the effect of mild, moderate, and severe hepatic impairment on PK, safety, and tolerability of venglustat compared with normal hepatic function in male and female participants aged 18 to 79 years.

Study details include:

* The total study duration per participant will be up to 42 days, including up to 21 days for screening and approximately 21 days from institutionalization to the end of study (EOS).
* Institutionalization is mandatory until the activities on D5 have been completed.
* Each participant will receive a single dose of venglustat.
* For hepatically impaired participants there will be a screening visit, a multi-day institutionalization visit, and 7 site visits after D5 discharge, including the end of study (EOS) visit.
* For healthy volunteers there will be a screening visit, a multi-day institutionalization visit and 3 site visits after D5 discharge, including the end of study (EOS) visit.

DETAILED DESCRIPTION:
The duration of the study for a participant in any arm will be up to 42 days. The treatment and follow up periods will last for a combined total of approximately 20 days, while the screening period will be up to 3 weeks, but may be shorter on an individual basis.

Screening period: up to 3 weeks (Days -21 to -2).

Open-label treatment period with compulsory institutionalization (Days -1 to 5).

Follow up period lasting until approximately day 20 ± 2 days post administration. This will include 7 additional site visits (including the EOS visit) for hepatically impaired groups. The group with normal hepatic function will only need to return D6 and D7 for study visit after institutionalization is completed.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 79 years of age inclusive, at the time of signing the informed consent.
* Body weight between 50.0 and 115.0 kg, inclusive, if male; between 40.0 and 100 kg, inclusive, if female, and body mass index (BMI) within the range 18 to 40 kg/m2, inclusive, at screening.
* Contraception (with double contraception methods) for male and female participants; not pregnant or breastfeeding for female participants; no sperm donation for male participants.
* Female participants must refrain from donating ova/ovum.
* Capable of giving signed informed consent.

Participants with mild, moderate, and severe hepatic impairment

* Stable chronic liver disease assessed by medical history, physical examination, and laboratory values. Hepatic impairment will be assessed according to the Child-Pugh classification, using CPS (Mild hepatic impairment is defined as a total score ranging from 5 to 6, inclusive (CPS-A); Moderate hepatic impairment is defined as a total score ranging from 7 to 9, inclusive (CPS-B); and severe hepatic impairment is defined as a total score ranging from 10 to 15, inclusive (CPS-C).
* Laboratory parameters within the acceptable range for participants with hepatic impairment; however, serum creatinine should be strictly at or below the upper laboratory norm and eGFR should be >= 60 mL/min.

Participants with normal hepatic function

* Certified as healthy by a comprehensive clinical assessment (detailed medical history and complete physical examination).
* Laboratory parameters within the reference range for healthy participants.

Exclusion Criteria:

* Participant who had severe course of COVID-19 (i.e., hospitalization, extracorporeal membrane oxygenation, mechanically ventilated) within the past 8 weeks.
* History of current recreational drugs or alcohol abuse.
* Smoking more than 15 cigarettes or equivalent per day.
* Symptomatic postural hypotension, whatever the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in SBP ≥30 mmHg within 3 minutes when changing from supine to standing position at screening and Day 1.
* Blood donation within 2 months before inclusion.
* Positive result on drug or alcohol screen.
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the Investigator, contraindicates participation in the study.
* Any consumption of citrus fruits (grapefruit, orange, etc) or their juices within 5 days before inclusion).
* Any participant who cannot comply with the following study restrictions: refraining from drinking alcohol, tea, coffee, chocolate, quinine, or caffeine-containing beverages from 1 day before institutionalization and throughout the study duration; following a stable lifestyle with no intensive physical activity from 1 day prior to institutionalization throughout the study duration until after collection of the final PK sample.
* Positive result on anti-human immunodeficiency virus (HIV) or COVID-19 test.

Participants with mild, moderate, and severe hepatic impairment

* Hepatocellular carcinoma.
* Acute hepatitis.
* Uncontrolled or decompensated hepatic encephalopathy. Encephalopathy grade > 2.
* Any drug (within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication) which could impact by any mechanism of action, the pharmacokinetics of the investigational medicinal product, including moderate and strong CYP3A4 inhibitors or inducers.
* Any participant enrolled in or having participated in this or any other clinical study involving an IMP or in any other type of medical research according to applicable regulations within the past 14 days or 5 half-lives before screening, whichever is longer, per local regulations.

Participants with normal hepatic functions

* Any history or presence of clinically relevant hepatic or renal disease.
* Any medication (including St John's Wort) within 14 days before inclusion or within 5 times the elimination half-life or pharmacodynamic half-life of the medication, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days and any biologics (antibody or its derivatives) given within 4 months before inclusion.
* Current enrollment OR past participation in another investigational study in which an investigational intervention (eg, drug, vaccine, invasive device) was administered within the last 14 days or 5 half-lives days before screening, whichever is longer per local regulations.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Maximum venglustat plasma concentration observed (Cmax) | Baseline to Day 20
Area under the plasma concentration versus time curve extrapolated to infinity (AUC) | Baseline to Day 20

SECONDARY OUTCOMES:
Time to maximum venglustat plasma concentration (tmax) | Baseline to Day 20
Number of participants with adverse event (AE), treatment emergent adverse events (TEAEs), serious adverse events (SAEs) and adverse events of special interest (AESI) | Baseline to Day 20

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (6):
- United States (5):
  - Inland Empire Liver Foundation Site Number : 8400004, Rialto, California
  - Clinical Pharmacology of Miami Site Number : 8400002, Miami, Florida
  - Nucleus Network Site Number : 8400001, Saint Paul, Minnesota
  - Volunteer Research Group-NOCCR Site Number : 8400003, Knoxville, Tennessee
  - American Research Corporation Site Number : 8400005, San Antonio, Texas
- Investigational Site Number : 2760001, Kiel, Germany

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: POP16551 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25334&tenant=MT_SNY_9011